CLINICAL TRIAL: NCT03670940
Title: Effect of Bronchiectasis on Respiratory Functions, Exercise Capacity, Dyspnea Perception and Quality of Life in COPD Patients
Brief Title: Bronchiectasis Effect in COPD Patients
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof., Izmir Katip Celebi University
Other Study IDs: IKC
Record Dates: First submitted 2018-09-12; First posted 2018-09-14 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Bronchiectasis; Copd
MeSH Terms: conditions — Bronchiectasis; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD patients: COPD patients without bronchiectasis
- COPD and bronchiectasis patients: COPD patients with bronchiectasis

SUMMARY:
The etiology of bronchiectasis, known as permanent, abnormal, and localized development of bronchi, varies. However, most of them are responsible for infections during childhood. The prevalence of bronchiectasis is particularly high in advanced COPD patients. This phenomenon, called COPD-bronchiectasis overlap syndrome, affects the clinic of COPD patients negatively. In this study; bronchiectasis in respiratory function, exercise capacity, dyspnoea and quality of life in COPD patients.

DETAILED DESCRIPTION:
The etiology of bronchiectasis, known as permanent, abnormal, and localized development of bronchi, varies. However, most of them are responsible for infections during childhood. The prevalence of bronchiectasis is particularly high in advanced COPD patients. This phenomenon, called COPD-bronchiectasis overlap syndrome, affects the clinic of COPD patients negatively. In this study; bronchiectasis in respiratory function, exercise capacity, dyspnoea and quality of life in COPD patients.

Torax CTs of patients with COPD who are admitted to the outpatient clinic will be examined. There will be two groups, group 1 in patients with COPD accompanied by bronchiectasis and group 2 in COPD patients without bronchiectasis. In both groups, respiratory function tests, exercise capacities, dyspnea perceptions and quality of life will be evaluated. The data will be compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old
* clinically stable

Exclusion Criteria:

* other respiratory disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with and without bronchiectasis.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 15 minutes
  six minute walk test

SECONDARY OUTCOMES:
Dyspnea Severity | 5 minutes
  mMRC Dyspnea Scale (0: no dyspnea, 4: very severe dyspnea)
Lung Function | 20 minutes
  Respiratory Function Test
Health Related Quality of Life | 25 minutes
  St. George Respiratory Questionnaire (maximum score: 100, lower score means better quality of life)

IPD SHARING:
Plan to Share IPD: No